CLINICAL TRIAL: NCT03115086
Title: A Prospective, Observational, Non-Interventional, Post-Marketing, Patient Registry to Collect Data on Routine Clinical Care in Patients Treated With Cholbam® (Cholic Acid)
Brief Title: The REPLACE Registry for Cholbam® (Cholic Acid)
Status: Active, not recruiting | Type: Observational
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 031CHO15001
Record Dates: First submitted 2017-01-10; First posted 2017-04-14 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Bile Acid Synthesis Disorders
Keywords: Bile Acid Synthesis Disorder; Zellweger Spectrum Disorder; Peroxisomal Disorder; Cholic Acid; Cholbam; The REPLACE Registry
MeSH Terms: conditions — Zellweger Syndrome; Peroxisomal Disorders | interventions — Cholic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Existing User: Patients who have been using Cholbam for at least 30 days
  Interventions: Drug: Cholbam
- New User: First-time initiators of Cholbam
  Interventions: Drug: Cholbam

INTERVENTIONS:
Drug: Cholbam — Cholbam prescribed according to the approved label.

SUMMARY:
This is a prospective, observational, non-interventional patient registry study designed to document product safety and effectiveness outcomes for 10 years in patients treated with Cholbam, including those who have been using Cholbam for at least 30 days (existing users) and those who are first-time initiators of Cholbam.

DETAILED DESCRIPTION:
No experimental intervention is involved. Patients in the Registry undergo clinical assessments and receive care as determined by the patient's treating physician.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients, of any age.
2. The patient and/or the patient's parent/legal guardian is willing and able to provide signed informed consent, and the patient, if less than 18 years of age, is willing to provide assent as appropriate and in accordance with local regulatory, IRB, and EC requirements.
3. The patient has a diagnosis for which Cholbam is indicated.
4. The patient is or will be treated with Cholbam at the time of signing the informed consent form (ICF) (enrollment).

Exclusion Criteria:

1. Patients who, by judgement of the Investigator, will not be able to comply with the requirements of the protocol will be excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with a diagnosis for which Cholbam is indicated are eligible for inclusion in the Registry.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2017-07-10 (Actual); Primary Completion 2038-07 (Estimated); Study Completion 2039-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with worsening cholestasis | 10 Years
  Worsening cholestasis will be identified by measuring direct total bilirubin concentration in blood and will be defined as a 25% increase from previous measurement if the total bilirubin is >1mg/dL.
Number of participants with new-onset cholestasis | 10 Years
  Patients with new-onset cholestasis will be identified by detecting abnormal direct bilirubin concentration >1mg/dL or direct bilirubin greater than 20% of the total bilirubin if total bilirubin is >5mg/dL.
Number of participants with steatorrhea leading to poor growth | 10 Years
  Steatorrhea leading to poor growth in children, which will be defined as a decrease in growth percentiles from the original percentile at enrollment to the registry study.
Changes in serum levels of fat-soluble vitamins | 10 Years
  Fat-soluble vitamin (A, D, E, K) deficiencies will be identified by comparing results from serum assays (Vitamin A: Retinol, Vitamin D: 250HD2 + 250HD3, Vitamin K: Serum Vitamin K, Vitamin E: Serum Vitamin E) for each vitamin with standard ranges.
Neuropathic signs or symptoms related to fat-soluble vitamin deficiencies | 10 Years
  Neuropathic signs or symptoms related to fat-soluble vitamin deficiencies (peripheral neuropathy, cerebellar ataxia) will be assessed by the Investigator.
Number of participants with growth failure | 10 Years
  Growth failure that the physician judges to be attributable to malabsorption.
Death | 10 Years
  AEs and SAEs leading to death will be recorded. The relatedness of death to Cholbam or disease progression will be recorded.
Adverse effects on pregnancy, pregnancy outcomes, and infant status | 10 Years
  Adverse effects on pregnancy, pregnancy outcomes, and infant status will be recorded.
All Adverse Events (AEs) and Serious AEs (SAEs) | 10 years
  All other AEs and SAEs will be collected.

SECONDARY OUTCOMES:
Changes in Cholbam dosing regimens and reasons for any dose modifications or treatment discontinuations | 10 years
Changes from baseline in weight | 10 years
  For patients aged 18 years of or less, these data will be converted into Z-scores based on the WHO growth standards for infants aged 0-2 years and the Centers for Disease Control and Prevention growth standards for children 2-20 years. Growth failure will be defined as a decrease in percentiles from the original percentile at entry point into the registry study.
Changes from baseline in length/height | 10 years
  For patients aged 18 years of or less, these data will be converted into Z-scores based on the WHO growth standards for infants aged 0-2 years and the Centers for Disease Control and Prevention growth standards for children 2-20 years. Some patients will be adult or will have achieved final height. Growth failure will be defined as a decrease in percentiles from the original percentile at entry point into the registry study.
Changes from baseline in head circumference in infants | 10 years
  For patients aged 18 years of or less, these data will be converted into Z-scores based on the WHO growth standards for infants aged 0-2 years and the Centers for Disease Control and Prevention growth standards for children 2-20 years. Growth failure will be defined as a decrease in percentiles from the original percentile at entry point into the registry study.
Age-appropriate developmental milestones in infants | 10 years
  Measured by WHO Motor Development Milestones
Changes in prothrombin time (PT) | 10 years
Changes in international normalized ratio (INR) | 10 years
Changes in albumin | 10 years
Changes in bilirubin | 10 years
Changes in direct bilirubin | 10 years
Changes in alanine aminotransferase (ALT) | 10 years
Changes in aspartate aminotransferase (AST) | 10 years
Changes in gamma-glutamyl transferase (GGT) | 10 years
Changes in alkaline phosphatase | 10 years
Presence or absence of urinary bile acids and levels of bile acid intermediaries and urinary bile alcohol | 10 years
All indications for which Cholbam has been prescribed | 10 years
  Description of all indications for which Cholbam has been prescribed

CONTACTS AND LOCATIONS:
Overall Officials: Sagar A Vaidya, MD, PhD, Study Director — Vice President, Clinical Development
Locations (23):
- United States (23):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Stanford School of Medicine, Palo Alto, California
  - UC San Francisco, San Francisco, California
  - Kidz Pediatric Multispecialty Group, Hollywood, Florida
  - Nemours duPont Pediatrics Specialty Clinic, Jacksonville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Children's Center For Digestive Health, Atlanta, Georgia
  - The Community Health Clinic, Topeka, Indiana
  - Ochsner Hospital for Children, New Orleans, Louisiana
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Office of Dr. Esperanza Font-Montgomery MD, Columbia, Missouri
  - Washington University at St Louis, St Louis, Missouri
  - Icahn School Of Medicine at Mount Sinai, New York, New York
  - Montefiore Medical Center, New York, New York
  - Golisano Children's Hospital, URMC, Rochester, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Monroe-Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Primary Children's Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No